CLINICAL TRIAL: NCT02006498
Title: A Randomised, Double-blind, Placebo-controlled, Phase II, Single-centre Study to Assess the Safety and Efficacy of Silymarin 700 mg Capsules TID for the Treatment of Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Silymarin for the Treatment of Non-Alcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Rottapharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LE13T0.01
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: non-alcoholic fatty liver disease; sillymarin; randomised trial; non-alcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Silymarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sillymarin (Experimental): Active component study medication
  Interventions: Drug: Sillymarin
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sillymarin — Sillymarin is derived from the milk thistle plant, Silybum marianum, a herbal remedy that has been used for centuries for diseases of the liver. It is a complex mixture of 6 major flavonolignans (silybins A and B, isosilybins A and B, silychristin, and silydianin), as well as other minor polyphenolic compounds.
  Other Names: Legalon
  Arms: Sillymarin
Drug: Placebo — Placebo capsule with same appearances as study drug
  Arms: Placebo

SUMMARY:
This is a randomised study to examine whether high dose Sillymarin will be able to help improve fat-induced liver damage in the liver. The study hypothesis is that high dose Sillymarin will be able to reduce steato-hepatitis (fat-related liver inflammation) better than placebo.

DETAILED DESCRIPTION:
OBJECTIVES OF STUDY Primary Objectives

1. To assess the safety and adverse event profile of Silymarin compared to placebo.
2. To assess the efficacy of Silymarin as defined by an improvement in non-alcoholic steatosis (NAS) activity score by at least 30% from baseline compared to placebo.

Secondary Objectives

1. To compare NAS activity before and after Silymarin therapy.
2. To characterize changes in ALT and AST during Silymarin therapy.
3. To compare insulin resistance measured by HOMAr during Silymarin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older.
* Diagnosed with NASH (refer to Section 5.2)
* AST and/or ALT greater than 40 IU/L.
* Must agree to adhere to alcohol consumption guideline.
* Weight gain//loss of no more than 10% between biopsy and screening or within 30 days of screening if the biopsy is performed during the screening period.
* No change in diabetic and/or lipid medications between biopsy and screening or within 30 days of screening if the biopsy is performed during the screening period

Exclusion Criteria:

* Use of silymarin or other milk thistle preparations for a period of 90 consecutive days or longer between biopsy and initial screening, or within 30 days prior to screening if the biopsy is performed during the screening period.

  * Use of other antioxidants or non-prescribed complementary alternative medications for a period of 90 consecutive days or longer between biopsy and initial screening, or within 30 days prior to screening if the biopsy is performed during the screening period.
  * Use of warfarin, metronidazole, or acetaminophen (greater than 2 grams per day) between screening and randomization.
  * Use of oral steroids for more than 14 days of screening or prior to randomization.
  * BMI ≥ 35 kg/m2 between screening and randomization.
  * Poorly-controlled diabetes (HbA1c > 8 %) between screening and randomization
  * Diabetes mellitus treated with oral agents other than the secretagogues or metformin between screening and randomization. Sitagliptin is allowed.
  * For patients using anti-hyperlipidemic agents or accepted anti-diabetic agents, any change of agent or dose between screening and randomization.
  * Radiologic imaging consistent with cirrhosis or portal hypertension.
  * Evidence of decompensated liver disease
  * Platelet count < 130 x 109 /L at screening.
  * History of bariatric surgery, or undergoing evaluation for bariatric surgery.
  * Known allergy/sensitivity to milk thistle or its preparations.
  * History of immunologically mediated disease
  * History of thyroid disease poorly controlled on prescribed medications.
  * History of solid organ or bone marrow transplantation.
  * Primary hepatic malignancy.
  * Secondary hepatic malignancy or extrahepatic malignancy.
  * Serum Creatinine of 176 μmol/L or greater or creatinine clearance (calculated according to Cockcroft-Gault) 60 mL/min or less, or on dialysis, at screening.
  * Severe illness or any other conditions that would make the patient, in the opinion of the investigator, unsuitable for the study.
  * Women with ongoing pregnancy or breast feeding, or contemplating pregnancy.
  * Women of childbearing potential who are not practicing an acceptable form of birth control.
  * Participation in a research drug trial within 30 days of screening.
  * Inability or unwillingness to give informed consent or abide by the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of Silymarin as defined by an improvement in non-alcoholic steatosis (NAS) activity score by at least 30% from baseline compared to placebo | 12 months

SECONDARY OUTCOMES:
To assess the safety and adverse event profile of Silymarin compared to placebo | 12 months

OTHER OUTCOMES:
To characterize changes in ALT and AST during Silymarin therapy | 12 months
To compare insulin resistance measured by HOMAr during Silymarin therapy. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Mahadeva, MD, MRCP, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Wah Kheong C, Nik Mustapha NR, Mahadeva S. A Randomized Trial of Silymarin for the Treatment of Nonalcoholic Steatohepatitis. Clin Gastroenterol Hepatol. 2017 Dec;15(12):1940-1949.e8. doi: 10.1016/j.cgh.2017.04.016. Epub 2017 Apr 15. PMID 28419855